CLINICAL TRIAL: NCT01393587
Title: A New Exogenous Marker for Diagnosis of Oxidative Stress During Laproscopic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Collaborators: Migal, Galilee Technology Center (Other)
Other Study IDs: BIC-2011
Record Dates: First submitted 2011-07-12; First posted 2011-07-13 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2011-07

CONDITIONS: Oxidative Stress; Laproscopy
Keywords: Oxidative Stress; Laproscopy

ARMS (1):
- Experimental (Experimental)
  Interventions: Procedure: Taking blood samples

INTERVENTIONS:
Procedure: Taking blood samples

SUMMARY:
Recently, a new synthetic marker was developed, based on a molecule that is composed of Amino Acids and Linoleic Acid and Neucleic Acid, which is capable of detecting even minor changes of oxidative stress.

The investigators would like to assess the usefulness of this marker during positive pressure pneumoperitoneum, during laproscopic surgery, with or without intenstinal resection (ischemia induced by intra-abdominal pressure and vascualr compromise).

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients undergoing elective laproscopic cholecystectomy and patients undergoing operation for tumer of large intenstine.

Exclusion Criteria:

* Patients suffering from Cardio Pulmonory and renal diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Western Galilee Hospital, Nahariya, Israel